CLINICAL TRIAL: NCT00871494
Title: A Multicenter, Non-Randomized, Open Label Study Of Azithromycin Intravenous Followed By Oral Administration In Japanese Adult Subjects With Pelvic Inflammatory Disease (PID) Requiring Initial Intravenous Therapy
Brief Title: Study Of Azithromycin Intravenous Formulation Against Pelvic Inflammatory Disease (PID) In Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661192
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-09

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin switch therapy (switch from intravenous to oral). (Experimental)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — The patients will receive 500 mg intravenous azithromycin QD for 1 to 2 days. The period of administration of intravenous dosing is judged by investigators according to patient status. Following intravenous administration, the patients will be received the 250 mg oral azithromycin (tablet formulation) QD to complete a total of 7 days therapy.

SUMMARY:
Azithromycin had a potent in vitro activities and broad spectrum from typical and atypical bacteria to anaerobes. Azithromycin intravenous formulation demonstrated high efficacy and eradication rate in the western clinical trials. Development of azithromycin intravenous formulation would bring the clinical benefit to patients with pelvic inflammatory disease (PID) in Japan.

ELIGIBILITY:
Inclusion Criteria:

Both of following symptoms should be observed.

* Lower abdominal pain and/or lower abdominal tenderness.
* Hypochondrial pain and/or hypochondrial tenderness (tenderness of uterus or adnexa of uterus).

Exclusion Criteria:

Known or suspected hypersensitivity or intolerance to azithromycin, other macrolides, or ketolides.

Hepatic dysfunction (AST, ALT, total bilirubin > 3 times institutional normal).

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- Japan (31):
  - Pfizer Investigational Site, Aichi-gun, Aichi-ken
  - Pfizer Investigational Site, Ichinomiya, Aichi-ken
  - Pfizer Investigational Site, Nagoya-city Naka-ku, Aichi-ken
  - Pfizer Investigational Site, Tanba-gun Fusou-chou, Aichi-ken
  - Pfizer Investigational Site, Hirosaki, Aomori
  - Pfizer Investigational Site, Niihama, Ehime
  - Pfizer Investigational Site, Kasuga, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Kitakyushu-shi, Yahatanishi-ku, Fukuoka
  - Pfizer Investigational Site, Chuou-ku, Fukuoka-city
  - Pfizer Investigational Site, Fukushima, Fukushima
  - Pfizer Investigational Site, Takasaki, Gunma
  - Pfizer Investigational Site, Takasaki-shi, Gunma
  - Pfizer Investigational Site, Hakodate-shi Goryoukaku-cho, Hokkaido
  - Pfizer Investigational Site, Hakodate-shi Hon-cho, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Chuo-ku, Hyōgo
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Kounoike Shinmachi, Kagoshima-city
  - Pfizer Investigational Site, Kagoshima, Kagoshima-ken
  - Pfizer Investigational Site, Kamigyou-ku, Kyoto-city
  - Pfizer Investigational Site, Nagano, Nagano
  - Pfizer Investigational Site, Suzaka-shi, Nagano
  - Pfizer Investigational Site, Okayama, Okayama-city
  - Pfizer Investigational Site, Okayama, Okayama-ken
  - Pfizer Investigational Site, Koshigaya, Saitama
  - Pfizer Investigational Site, Aoba-ku, Sendai-city
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Nakaku, Yokohama-city Kanagawa
  - Pfizer Investigational Site, Fukushima

REFERENCES:
- [Derived] Mikamo H, Iwasaku K, Yamagishi Y, Matsumizu M, Nagashima M. Efficacy and safety of intravenous azithromycin followed by oral azithromycin for the treatment of acute pelvic inflammatory disease and perihepatitis in Japanese women. J Infect Chemother. 2014 Jul;20(7):429-35. doi: 10.1016/j.jiac.2014.04.001. Epub 2014 Apr 29. PMID 24787738
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661192&StudyName=Study%20Of%20Azithromycin%20Intravenous%20Formulation%20Against%20Pelvic%20Inflammatory%20Disease%20%28PID%29%20In%20Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: Azithromycin switch therapy (from 500 mg intravenous azithromycin once daily for 1 to 2 days to 250 mg oral azithromycin once daily to complete a total of 7 days therapy)
Period: Overall Study
Arm/Group | Azithromycin
Started | 76
Completed | 62
Not Completed | 14
Not completed — Protocol Violation | 5
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Azithromycin
Number analyzed (Participants) | 76
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Clinical Response, Data Review Committee Assessment) in Participants Who Enrolled After Protocol Amendment (the Inclusion Criterion Regarding Fever of 37℃ or Higher Was Option)
Description: Response rate was calculated from the following formula, "the number of participants assessed as effective" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
  The inclusion criterion regarding fever was amended from the required criteria to the additional criteria in consultation with the regulatory authority. The subset of participants who were enrolled after the protocol amendment was the primary analysis sets for efficacy.
Time Frame: End of Treatment, Day 15 and Day 29
Population: Clinical per protocol set consisted of all participants who received at least one dose, had no significant violation of protocol, and underwent prescribed evaluations during the observation period. No imputation was used for missing data. "n" in the Measure Categories means total participants excluding ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 51
percentage of participants
  End of Treatment (n=51) | 94.1 [83.8 to 98.8]
  Day 15 (n=51) | 94.1 [83.8 to 98.8]
  Day 29 (n=46) | 93.5 [82.1 to 98.6]

2. Secondary Outcome: Response Rate (Clinical Response, Investigator Assessment) in Participants Who Enrolled After Protocol Amendment (the Inclusion Criterion Regarding Fever of 37℃ or Higher Was Option)
Description: as for outcome 1
Time Frame: End of Treatment, Day 15 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 51
percentage of participants
  End of Treatment (n=51) | 92.2 [81.1 to 97.8]
  Day 15 (n=48) | 100 [92.6 to 100]
  Day 29 (n=46) | 100 [92.3 to 100]

3. Secondary Outcome: Eradication Rate (Bacteriological Response, Data Review Committee Assessment) in Participants Who Enrolled After Protocol Amendment (the Inclusion Criterion Regarding Fever of 37℃ or Higher Was Option)
Description: Eradication Rate was calculated from the following formula, "the number of participants assessed as eradication, presumed eradication and microbial substitution" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
  The inclusion criterion regarding fever was amended from the required criteria to the additional criteria in consultation with the regulatory authority. The subset of participants who were enrolled after the protocol amendment was the primary analysis sets for efficacy.
Time Frame: End of treatment, Day 15, Day 29
Population: Bacteriologic per protocol set consisted of all participants in the clinical per protocol set in whom bacterial pathogens were identified at baseline. No imputation was used for missing data. "n" in the Measure Categories was the total participants EXCLUDING ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 36
percentage of participants
  End of treatment (n=31) | 77.4 [58.9 to 90.4]
  Day 15 (n=34) | 85.3 [68.9 to 95.0]
  Day 29 (n=31) | 83.9 [66.3 to 94.5]

4. Secondary Outcome: Eradication Rate (Bacteriological Response, Investigator Assessment) in Participants Who Enrolled After Protocol Amendment (the Inclusion Criterion Regarding Fever of 37℃ or Higher Was Option)
Description: Eradication Rate was calculated from the following formula, "the number of participants assessed as eradication , presumed eradication and microbial substitution" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
  The inclusion criterion regarding fever was amended from the required criteria to the additional criteria in consultation with the regulatory authority. The subset of participants who were enrolled after the protocol amendment was the primary analysis sets for efficacy.
Time Frame: End of treatment, Day 15, Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentageof participants
Arm/Group | Azithromycin
Number analyzed (Participants) | 36
percentageof participants
  End of treatment (n=14) | 85.7 [57.2 to 98.2]
  Day 15 (n=11) | 85.7 [63.7 to 97.0]
  Day 29 (n=19) | 89.5 [66.9 to 98.7]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Azithromycin
Serious Adverse Events (participants affected / at risk) | 3/76
Other Adverse Events (participants affected / at risk) | 35/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=76)
Lymphadenitis (Blood and lymphatic system disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=76)
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 10
Gastritis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Injection site pain (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 4
Vaginitis bacterial (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Ovulation pain (Pregnancy, puerperium and perinatal conditions) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.